CLINICAL TRIAL: NCT04767152
Title: Clinical Study of the Therapy Neurotoxicity Using Quantitative Assessment of the Brain Structures and Functions by MRI, EEG and Evoked Potentials in Patients With Acute Lymphoblastic Leukemia Over 6 Years Old
Brief Title: Evaluation of Brain Changes in ALL Patients on Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCPHOI-2019-07
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Acute Leukemia
Keywords: Quantitative MRI; acute lymphoblastic leukemia; neurotoxity; children
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — The quantitative assessment of MRI parameters, The macromolecular proton fraction (MPF) (%) in brain tissue. Before the start of therapy - the starting point. Point 2. 36 ± 3 days after the start of the therapy. Point 3. After completing three courses of consolidation chemotherapy. Point 4. After confirmation of remission status, optionally provided.

SUMMARY:
The study is aimed at assessing changes in the brain of patients from 6 to 18 years old with a diagnosis of acute lymphoblastic leukemia during chemotherapy.

DETAILED DESCRIPTION:
Children with acute lymphoblastic leukemia receive long-term combined chemotherapy treatment, one of the main part of this treatment is methotrexate. Methotrexate can cause acute, subacute, and long-term neurotoxicity. Clinical symptoms of neurotoxicity, such as seizures, aphasia, are often associated with leukoencephalopathy. However, leukoencephalopathy may develop asymptomatically in children receiving methotrexate.

The effect of chemotherapy on the neurological status of patients is widely covered in the literature. There are very few studies devoted to the quantitative assessment of MRI parameters, especially in children. MRI is a non-invasive method that does not harm the patient and can be used to assess absolutely all structures of the brain.

ELIGIBILITY:
Inclusion Criteria:

1. patients from 6 to 18 years old
2. diagnosis of acute lymphoblastic leukemia during chemotherapy

Exclusion Criteria:

1. patients less then 6, and older then 18 years old
2. patients who cannot perform the study MRI without general anesthesia
3. Refusal to sign informed consent.
4. The presence of absolute contraindications to MRI studies.
5. Extremely serious condition of the patient.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-21 (Estimated)

PRIMARY OUTCOMES:
percentage of the macromolecular proton fraction (MPF) in brain tissue. | Before the start of therapy
  macromolecular proton fraction (MPF) in brain tissue.
percentage of the macromolecular proton fraction (MPF) in brain tissue. | 36 ± 3 days after the start of the therapy..
  macromolecular proton fraction (MPF) in brain tissue.
percentage of the macromolecular proton fraction (MPF) in brain tissue. | ap to 1 week After completing three courses of consolidation chemotherapy.
  macromolecular proton fraction (MPF) in brain tissue.
percentage of the macromolecular proton fraction (MPF) in brain tissue. | ap to 1 week After confirmation of remission status, optionally provided.
  macromolecular proton fraction (MPF) in brain tissue.

SECONDARY OUTCOMES:
T1 maping | Point 1. Before the start of therapy - the starting point. Point 2. 36 ± 3 days after the start of the therapy. Point 3. 4 mounths ± 1 week after the start of the therapy. Point 4. through study completion, an average of 2 year
  T1 mapping (ms) is a magnetic resonance imaging technique used to calculate at 4 time points
apparent diffusion coefficient | Point 1. Before the start of therapy - the starting point. Point 2. 36 ± 3 days after the start of the therapy. Point 3. 4 mounths ± 1 week after the start of the therapy. Point 4. through study completion, an average of 2 year
  value of apparent diffusion coefficient in mm2/s calculated at 4 time points
percentage of the water myelin fraction | Point 1. Before the start of therapy - the starting point. Point 2. 36 ± 3 days after the start of the therapy. Point 3. 4 mounths ± 1 week after the start of the therapy. Point 4. through study completion, an average of 2 year
  water myelin fraction calculated at 4 time points
value of the cerebral blood flow | Point 1. Before the start of therapy - the starting point. Point 2. 36 ± 3 days after the start of the therapy. Point 3. 4 mounths ± 1 week after the start of the therapy. Point 4. through study completion, an average of 2 year
  cerebral blood flow (CBF) (ml/100g/min) in brain tissue. calculated at 4 time points

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev Federal Research and Clinical Centre of Paediatric Haematology, Oncology and Immunology, Moscow, Russia